CLINICAL TRIAL: NCT03504813
Title: Technologies for Participatory Medicine and Health Promotion in the Elderly Population
Acronym: GERIATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Geriatros (Other); Center on Information and Communication Technologies (Other); Instituto de Investigacion Biomedica de A Coruna (Other); Aldaba (Unknown); Cobián Clinic (Unknown)
Responsible Party: Principal Investigator, Javier Pereira, Proffesor PhD, Universidade da Coruña
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IN852A 2016/10
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Aging; Age Problem
Keywords: Elderly; Quality of life; Wearables; Urinary incontinence; Insomnia; Risk of falls
MeSH Terms: conditions — Urinary Incontinence; Sleep Initiation and Maintenance Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Urinary Incontinence (Experimental): The involuntary loss of urine through the urethra, objectively demonstrable and constituting for the person who suffers it a social and hygienic problem.
  In this arm, participants will receive the following interventions: physical activities program, training of the pelvic floor and counseling about occupational performance
  Interventions: Other: Physical activities program; Other: Training of the pelvic floor; Behavioral: Counseling about occupational performance
- Insomnia (Experimental): A condition characterized by an unsatisfactory amount or quality of sleep which persists for a considerable period. This disorder includes difficulties for the falling and/or staying asleep and early awakening in the final phase of sleep.
  In this arm, participants will receive the following interventions: physical activities program, relaxation training and counseling about occupational performance.
  Interventions: Other: Physical activities program; Other: Relaxation training; Behavioral: Counseling about occupational performance
- Risk of falls (Experimental): Involuntary events that cause people to lose balance and find themselves on the ground or other firm surfaces. The factor of falls can be intrinsic (related to the person) or extrinsic (derived from the activity or environment of the individual).
  In this arm, participants will receive the following interventions: physical activities program, and counseling about occupational performance
  Interventions: Other: Physical activities program; Behavioral: Counseling about occupational performance

INTERVENTIONS:
Other: Physical activities program — To implement this line, the protocol of the VIVIFRAIL Project will be used as a reference. That protocol has different physical exercises, divided into itineraries, in order to adapt it to a person's capability. Several sessions of this research line will employ the use of videogames so that the elderly can explore new forms of physical activity and thus establish contact and expertise with new technologies. It is estimated that two sessions per week over two months are needed for each person to continue doing physical activity independently and with autonomy.
Other: Relaxation training — Will take place with those participants who are included in the research lines of insomnia and risk of falls. It is estimated that two sessions per week for one month are needed.
  Arms: Insomnia
Other: Training of the pelvic floor — the intervention will apply to participants enrolled in the research line dealing with urinary incontinence during the six months of intervention, with a frequency of two sessions per week
  Arms: Urinary Incontinence
Behavioral: Counseling about occupational performance — After the physical activity and relaxation programs, the counselling will start. With each participant, routines and daily activities will be planned that will be adequate according to different recommendations about urinary incontinence, insomnia and risk of falls. Different performance guidelines will be established in order to establish a good balance between activities. The guidelines can include the recommendations about adjustments to the environment. It is estimated that three sessions per week for two months are needed to incorporate advice and routines into the daily lives of participants.

SUMMARY:
Introduction: The progressive aging of the population is a socio-demographic phenomenon experienced by most countries in the world in recent decades, especially in Japan and in many European Union countries. During this process, so-called "geriatric syndromes" frequently occur. The focus of this study is the quality of life of the elderly in relation to these three factors: risk of falls, urinary incontinence, and insomnia.

Objective: The main purpose is to determine the impact of a multifactorial intervention program implemented with institutionalized elderly people. The program is focused on the treatment of the aforementioned factors.

Methods and Analysis: The study will be carried out with elderly people living in three residences for the elderly in A Coruña Province (Galicia, Spain).

It is a prospective and longitudinal study, with a temporary series design of a "quasi-experimental" type that evaluates the effect of an intervention in one given population by doing assessments pre- and post-intervention, but there is no comparison with a control group.

The intervention will be based on a multifactorial program, including the following phases: the use of wearable devices (wearable fitness trackers to register physical activity and sleep), the use of an App on a Tablet to record the participants' occupations and activities, counseling about performance in activities of daily living, the implementation of a physical activity program, and the treatment of the pelvic floor (according to each research line). The Quality of Life (QoL) will be assessed before and after the intervention, with the use of the questionnaire EuroQol-5D-5L. Data analysis will be applied with all registered variables through a quantitative perspective.

ELIGIBILITY:
Inclusion Criteria:

* People 65 years of age or older.

Specific criteria for each research line:

* Urinary incontinence:

  1. To have stress, urgency or mixed urinary incontinence
  2. To be a woman
* Insomnia:

  a) Diagnosis of insomnia and/or hypersomnia.
* Risk of falls:

  1. To have a previous history of falls in the last 6-12 months.
  2. To present risk of falling and/or fear of falling.
  3. To have independence in locomotion.

Exclusion Criteria:

* Showing cognitive deterioration from moderate to very severe (Mini-Examination Cognitive minor of 20 points).
* Having severe, acute complications in health that prevent assiduity in attending interventions.
* Diagnosis of conditions and/or pathologies in which physical activity is contraindicated (mainly cardiorespiratory diseases).
* Being in the final stage of a terminal illness.
* Bing in a situation of request for transfer to another center.
* Having a temporary stay in elderly residence.
* Having a situation of legal incapacity.

For the research line on urinary incontinence, several specific exclusion criteria have been established:

* Having functional urinary incontinence because that type is related to cognitive deterioration, urinary infection, polypharmacy, psychological problems, endocrinopathy, mobility restriction, and fecal incontinence.
* Having undergone surgery in the pelvic floor area.
* Uterine prolapse, cystocele and/or rectocele (levels 3-4).
* No control of the pelvic floor.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — One of interventions that are carrying on in the present study, is focused in prevention and treatment the urinary incontinence. For that, a pelvic floor training is implementing. For that, specific inclusion criteria has been established: the training is doing with a sample of women older than 65 years old.
Enrollment: 57 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the quality of life | Baseline and 6 months later (during intervention). Three months after intervention
  The variable will be determined with EuroQol-5D-5L. This descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

SECONDARY OUTCOMES:
Independence on Activities of Daily Living | Baseline and 6 months later (during intervention). Three months after intervention
  Barthel Activities of Daily Living (ADL) Index: This tool is used as a simple index of independence to score the ability of a patient to care for himself, and by repeating the test periodically, to assess his improvement. The performance is assessed based on these scores: <20: total dependence, 20---40: severe dependence, 45-55: moderate dependence, and 60 or more: mild dependence.
Gait and balance | Baseline and 6 months later (during intervention). Three months after intervention
  The test is scored on the individual's ability to perform specific tasks. "Scoring of the Tinetti Assessment Tool is done on a three-point ordinal scale with a range of 0 to 2. A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score (12 points), an overall balance assessment score (16 points), and a combined gait and balance score (28).
Cognitive State | Baseline and 6 months later (during intervention). Three months after intervention
  Mini-Mental State Examination (MMSE): This tool has been designed to determine the "cognitive state," that is one of the study's variables. It presents six values: one for each section (Orientation, Fixation, Concentration and calculation, Memory and Language, and Construction)
Oxford Grading Scale | Baseline and 3 months after intervention
  This scale measures the variable of "pelvic floor contractile capacity". It has a unique numerical value (0-5), that is the result from assessment of the contractile capacity of the pelvic floor muscles
Sandvick Severity Index | Baseline and 3 months after intervention
  This test assesses the variable "urine leakage". It presents a unique numerical value and consists of two questions, one of them about the frequency with which a person has urine leakage (maximum score of 4 points) and another with reference to the amount of urine in the exhaust (maximum score of 3 points)
24-Hour Pad Test | Baseline and 6 months later (during intervention). Three months after intervention
  This tool allows to measure the "amount of urine". This scale has three values (net weight of the napkin/diaper, weight with urine and weight difference).
Pelvic Floor Muscle Assessment: PERFECT Scheme | Baseline and 6 months later (during intervention). Three months after intervention
  The tool PERFECT Scheme allows to assess the "pelvic floor musculature". PERFECT is an acronym with P representing power (or pressure, a measure of strength using a manometric perineometer), E = endurance, R = repetitions, F = fast contractions, and ECT = every contraction timed.
International Consultation on Incontinence Questionnaire (Short Form) | Baseline and 6 months later (during intervention). Three months after intervention
  Self-administered questionnaire that qualifies the "symptoms and quality of life" in both male and female adult patients with symptoms of urine loss. It has 6 items, Score is 0 - 21 with a higher score indicating greater severity.
Oviedo Sleep Questionnaire | Baseline and 6 months later (during intervention). Three months after intervention
  This scale allows assess the "sleep satisfaction". It consists of 13 items with three values: one for each section (sleep satisfaction, insomnia and hypersomnia). Each item is scored from 1 to 5, except for item 1 which is scored from 1 to 7. The subscale of insomnia ranges from 9 to 45 points; the higher the score the greater the severity.
Pittsburgh Sleep Quality Assessment | Baseline and 6 months later (during intervention). Three months after intervention
  The measure consists of 19 individual items, creating seven components that produce one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Timed Get Up and Go Test | Baseline and 6 months later (during intervention). Three months after intervention
  A simple test used to assess a person's mobility and requires both static and dynamic balance
Falls Efficacy Scale International | Baseline and 6 months later (during intervention). Three months after intervention
  The tool measures "the level of concern about falling" during social and physical activities inside and outside the home. Individuals are asked to rate, on a four-point Likert scale,their concerns aboutthe possibility offalling when performing 16 activities.The scores are added up to calculate a total score that ranges from 16 to 64 for the FES-I and 8 to 28 for the short FES-I. A higher score indicates a greater fear of falls

OTHER OUTCOMES:
Charlson Comorbidity Index | 1 month before intervention
  Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
Incontinence Urinary-4 Questionnaire | 1 month before intervention
  This tool helps to classify the type of urinary incontinence (UI). This scale has a unique qualitative value (four different options). It is emphasized that question 1 identifies the effort of UI, while questions 2 and 3 identify the UI of urgency. Each question is answered as yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Javier P Pereira, PhD, Principal Investigator — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Gershenfeld N, Krikorian R, Cohen D. The Internet of things. Sci Am. 2004 Oct;291(4):76-81. doi: 10.1038/scientificamerican1004-76. No abstract available. PMID 15487673
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krle A-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 Statement: defining standard protocol items for clinical trials. Rev Panam Salud Publica. 2015 Dec;38(6):506-14. PMID 27440100
- [Background] Davies A, De Souza LH, Frank AO. Changes in the quality of life in severely disabled people following provision of powered indoor/outdoor chairs. Disabil Rehabil. 2003 Mar 18;25(6):286-90. doi: 10.1080/0963828021000043734. PMID 12623619
- [Background] Stier-Jarmer M, Grill E, Muller M, Strobl R, Quittan M, Stucki G. Validation of the comprehensive ICF Core Set for patients in geriatric post-acute rehabilitation facilities. J Rehabil Med. 2011 Jan;43(2):102-12. doi: 10.2340/16501977-0617. PMID 21042699
- [Background] Wade DT, Collin C. The Barthel ADL Index: a standard measure of physical disability? Int Disabil Stud. 1988;10(2):64-7. doi: 10.3109/09638288809164105. PMID 3042746
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Ferreira CH, Barbosa PB, de Oliveira Souza F, Antonio FI, Franco MM, Bo K. Inter-rater reliability study of the modified Oxford Grading Scale and the Peritron manometer. Physiotherapy. 2011 Jun;97(2):132-8. doi: 10.1016/j.physio.2010.06.007. Epub 2010 Oct 22. PMID 21497247
- [Background] Sandvik H, Seim A, Vanvik A, Hunskaar S. A severity index for epidemiological surveys of female urinary incontinence: comparison with 48-hour pad-weighing tests. Neurourol Urodyn. 2000;19(2):137-45. doi: 10.1002/(sici)1520-6777(2000)19:23.0.co;2-g. PMID 10679830
- [Background] Badia Llach X, Castro Diaz D, Perales Cabanas L, Pena Outerino JM, Martinez-Agullo E, Conejero Sugranes J, Arano Beltran P, Marques Queimadelos A, Roset Gamisans M, Perulero Escobar N. [The development and preliminary validation of the IU-4 questionnaire for the clinical classification of urinary incontinence]. Actas Urol Esp. 1999 Jul-Aug;23(7):565-72. Spanish. PMID 10488609
- [Background] Krhut J, Zachoval R, Smith PP, Rosier PF, Valansky L, Martan A, Zvara P. Pad weight testing in the evaluation of urinary incontinence. Neurourol Urodyn. 2014 Jun;33(5):507-10. doi: 10.1002/nau.22436. Epub 2013 Jun 24. PMID 23797972
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Derived] Nieto-Riveiro L, Groba B, Miranda MC, Concheiro P, Pazos A, Pousada T, Pereira J. Technologies for participatory medicine and health promotion in the elderly population. Medicine (Baltimore). 2018 May;97(20):e10791. doi: 10.1097/MD.0000000000010791. PMID 29768372
- See also: Barry A, McGwire S PK. Global AgeWatch Index 2015 [Internet]. Age International, editor. 2015 — https://fiapam.org/wp-content/uploads/2015/09/helpage-indice-global-envejecimiento-2015.pdf
- See also: Instituto Nacional de Estadistica. (Spanish Statistical Office) — http://www.ine.es/
- See also: World Health Organization. ICD-10 Version:2008 [Internet]. WHO, editor. Genebra; 2008 — https://www.who.int/classifications/icd/icdonlineversions/en/
- See also: World Health Orgnization. WHO | Falls [Internet]. WHO. World Health Organization; 2018 — http://www.who.int/mediacentre/factsheets/fs344/en/
- See also: Alberich T, Barranco Carrillo A, Funes Jiménez E, Espadas Alcázar MA, Melón González O. Intervención social y sanitaria con mayores manual para el trabajo con la 3a. y 4a. edad. — https://dialnet.unirioja.es/servlet/articulo?codigo=2706553
- See also: Millán Calenti JC. Gerontología y geriatría : valoración e intervención [Internet]. Editorial Médica Panamericana; 2011 — https://www.medicapanamericana.com/Libros/Libro/4308/Gerontologia-y-Geriatria.html
- See also: Giner P, Cetina C, Fons J, Pelechano V. Developing Mobile Workflow Support in the Internet of Things — http://lbd.udc.es/jornadas2011/actas/JISBD/JISBD/S7/YaPublicados/resumen_jisbd2011camerareadyColaborativos.pdf
- See also: Aceytuno M, Ascensión E, Miralles R, Prado B, Riera M, Roqueta C et al. Guía de buena práctica clínica en Geriatría. Incontinencia urinaria [Internet]. SEGG, editor. Barcelona; 2008 — https://www.segg.es/media/descargas/Acreditacion%20de%20Calidad%20SEGG/CentrosDia/GBPCG%20INCONTINENCIA%20URINARIA.pdf
- See also: Universidad Pública de Navarra. ViviFrail — http://www.vivifrail.com
- See also: Babes ' J, Gonllez ' MP, Vallejo J, S&z3 J, Gibert4 J, Ayuso5 JL, et al. S162 PI Affective disorders and antidepressants m] Oviedo Sleep Questionnaire (QSQ): — http://www.academia.edu/19465952/Oviedo_Sleep_Questionnaire_OSQ_A_new_semistructured_Interview_for_sleep_disorders

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03504813/Prot_SAP_000.pdf